CLINICAL TRIAL: NCT00732654
Title: The Safety and Efficacy of Sublingual/Oral Immunotherapy for the Treatment of Milk Protein Allergy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Duke University (Other); Greer Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00732654
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Milk Allergy
Keywords: Food Allergy; Oral Immunotherapy; Immunoglobulin E
MeSH Terms: conditions — Milk Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sublingual Immunotherapy (SLIT) (Experimental): These subjects will have a dose escalation of the milk protein extract given sublingually. After dose escalation, they will continue on the sublingual daily maintenance dose for approximately one year.
  Milk Protein Extract Immunotherapy : Sublingual extract daily in escalating doses to goal of 7mg/day for approximately 1 1/2 years.
  Interventions: Drug: Milk Protein Extract Immunotherapy goal of 4mg/day; Drug: Milk Protein Extract Immunotherapy goal of 7mg/day
- SLIT/ Oral Immunotherpay (OIT) B (Experimental): These subjects will start with a dose escalation of the milk protein extract given sublingually, and then will switch to milk powder given orally and will undergo a dose escalation for a goal of 1000 mg. After dose escalation, they will continue on the oral daily maintenance dose for approximately one year.
  Milk Powder Immunotherapy : Milk powder given orally in escalating doses with a goal of 1000mg/day for approximately 1 1/2 years.
  Interventions: Drug: Milk Protein Extract Immunotherapy goal of 4mg/day; Drug: Milk Powder Immunotherapy goal dose 1000mg/day
- SLIT/ OIT A (Experimental): These subjects will start with a dose escalation of the milk protein extract given sublingually, and then will switch to milk powder given orally and will undergo a dose escalation for a goal of 2000 mg. After dose escalation, they will continue on the oral daily maintenance dose for approximately one year.
  Milk Powder Immunotherapy : Milk powder given orally in escalating doses with a goal dose of 2000mg/day given for approximately 1 1/2 years.
  Milk Protein Extract Immunotherapy : Sublingual extract given daily in escalating doses with goal of 4 mg/day for approximately 20 weeks.
  Interventions: Drug: Milk Protein Extract Immunotherapy goal of 4mg/day; Drug: Milk Powder Immunotherapy goal dose 2000 mg/day

INTERVENTIONS:
Drug: Milk Protein Extract Immunotherapy goal of 4mg/day — Sublingual extract given daily in escalating doses with goal of 4 mg/day for approximately 20 weeks.
Drug: Milk Protein Extract Immunotherapy goal of 7mg/day — Sublingual extract daily in escalating doses to goal of 7mg/day for approximately 1 1/2 years.
  Arms: Sublingual Immunotherapy (SLIT)
Drug: Milk Powder Immunotherapy goal dose 2000 mg/day — Milk powder given orally in escalating doses with a goal dose of 2000mg/day given for approximately 1 1/2 years.
  Arms: SLIT/ OIT A
Drug: Milk Powder Immunotherapy goal dose 1000mg/day — Milk powder given orally in escalating doses with a goal of 1000mg/day for approximately 1 1/2 years.
  Arms: SLIT/ Oral Immunotherpay (OIT) B

SUMMARY:
The purpose of this study is to determine if small oral and sublingual doses of milk protein are safe and effective in decreasing sensitivity to cow's milk in allergic children.

ELIGIBILITY:
Inclusion Criteria:

* Are age 6 to 21 years
* Provide signed informed consent (by parent or legal guardian if the subject is a minor), and informed assent if applicable
* Have a history of symptomatic reactivity to cow's milk (i.e. Eczema, urticaria, upper or lower respiratory symptoms, GI disturbances, other rash or oral symptoms)
* Have a positive skin prick test (defined as wheal 3 mm ≥ negative control) and cow's milk- immunoglobulin E (IgE) > 0.35 kilo Immunoglobulin Units (kIU)/L
* Have a positive OFC to cow's milk at a cumulative dose of less than 184 milligrams of cow's milk intact protein (2,400 mg total milk protein).
* Are using appropriate birth control if subject is female and of child bearing age.
* Have self-injectable epinephrine (ie. EpiPen® or EpiPen Jr.®) available at home

Exclusion Criteria:

* Have a history of severe anaphylaxis defined as hypoxia (cyanosis or SpO2 ≤ 92% at any stage), hypotension, confusion, collapse, loss of consciousness; or incontinence
* Have a history of intubation related to asthma
* Tolerate more than 184 milligrams of intact cow's milk protein at initial OFC
* Are pregnant or lactating
* Have a viral Upper Respiratory Infection (URI) or gastroenteritis within 7 days of OFC (OFC needs to be rescheduled)
* Have pulmonary function tests <80% of predicted (FEV1) or clinical history consistent with more than moderate persistent asthma
* Are currently taking greater than medium dose inhaled corticosteroid (>400 mcg/day fluticasone or fluticasone equivalent if ≤ 12 years old or > 600 mcg/day if > 12 years old)
* Are unable to discontinue antihistamines for 5 days for long acting and 3 days for short acting prior to skin testing or food challenges
* Have used systemic corticosteroids within 4 weeks prior to baseline visit
* Are receiving omalizumab, beta-blocker, Angiotensin Converting Enzyome (ACE) inhibitor or tricyclic antidepressant therapy
* Have a chronic disease (other than asthma, atopic dermatitis or rhinitis) requiring therapy (e.g., heart disease, diabetes)
* Have participated in any interventional study for treatment of a food allergy in the past 12 months
* Have a severe reaction at initial DBPCFC, defined as either:

Life-threatening anaphylaxis, or Reaction requiring hospitalization

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2008-08; Primary Completion 2010-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Duke University, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 33 patients underwent screening Double-Blinded Placebo-Controlled Food Challenges (DBPCFCs). Two subjects failed screening because they tolerated at least 2.5g at the initial DBPCFC. One subject declined to continue in the study after the food challenge. 30 subjects were randomized.
Groups:
- SLIT: These subjects will have a dose escalation of the milk protein extract given sublingually. After dose escalation, they will continue on the sublingual daily maintenance dose for approximately one year.
  Milk Protein Extract Immunotherapy : Sublingual extract daily in escalating doses to goal of 7mg/day for approximately 1 1/2 years.
- SLIT/OIT B: These subjects will start with a dose escalation of the milk protein extract given sublingually, and then will switch to milk powder given orally and will undergo a dose escalation for a goal of 2000 mg. After dose escalation, they will continue on the oral daily maintenance dose for approximately one year.
  Milk Powder Immunotherapy : Milk powder given orally in escalating doses with a goal dose of 2000mg/day given for approximately 1 1/2 years.
  Milk Protein Extract Immunotherapy : Sublingual extract given daily in escalating doses with goal of 4 mg/day for approximately 20 weeks.
- SLIT/ OIT A: These subjects will start with a dose escalation of the milk protein extract given sublingually, and then will switch to milk powder given orally and will undergo a dose escalation for a goal of 1000 mg. After dose escalation, they will continue on the oral daily maintenance dose for approximately one year.
  Milk Powder Immunotherapy : Milk powder given orally in escalating doses with a goal of 1000mg/day for approximately 1 1/2 years.
  Milk Protein Extract Immunotherapy : Sublingual extract given daily in escalating doses with goal of 4 mg/day for approximately 20 weeks.
Period: Overall Study
Arm/Group | SLIT | SLIT/OIT B | SLIT/ OIT A
Started | 10 | 10 | 10
Completed | 10 | 9 | 10
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- OITA Group: These subjects will start with a dose escalation of the milk protein extract given sublingually, and then will switch to milk powder given orally and will undergo a dose escalation for a goal of 2000 mg. After dose escalation, they will continue on the oral daily maintenance dose for approximately one year.
  Milk Powder Immunotherapy : Milk powder given orally in escalating doses with a goal dose of 2000mg/day given for approximately 1 1/2 years.
  Milk Protein Extract Immunotherapy : Sublingual extract given daily in escalating doses with goal of 4 mg/day for approximately 20 weeks.
- OITB Group: These subjects will start with a dose escalation of the milk protein extract given sublingually, and then will switch to milk powder given orally and will undergo a dose escalation for a goal of 1000 mg. After dose escalation, they will continue on the oral daily maintenance dose for approximately one year.
  Milk Powder Immunotherapy : Milk powder given orally in escalating doses with a goal of 1000mg/day for approximately 1 1/2 years.
  Milk Protein Extract Immunotherapy : Sublingual extract given daily in escalating doses with goal of 4 mg/day for approximately 20 weeks.
- SLIT Group: These subjects will have a dose escalation of the milk protein extract given sublingually. After dose escalation, they will continue on the sublingual daily maintenance dose for approximately one year.
  Milk Protein Extract Immunotherapy : Sublingual extract daily in escalating doses to goal of 7mg/day for approximately 1 1/2 years.
- Total: Total of all reporting groups
Arm/Group | OITA Group | OITB Group | SLIT Group | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 10 | 10 | 30
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6 | 12
  Male | 7 | 7 | 4 | 18
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30
History of anaphylaxis to Cow's Milk (CM) [Count of Participants; unit: Participants] | 6 | 9 | 8 | 23
Other Food Allergies [Count of Participants; unit: Participants] | 6 | 8 | 9 | 23
Asthma [Count of Participants; unit: Participants] | 9 | 9 | 8 | 26
Atopic Dermatitis [Count of Participants; unit: Participants] | 6 | 6 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in CM-specific Immunogloblin E (IgE)
Description: Cow's milk specific IgE was measured at baseline and after therapy (kUa/L)
Time Frame: Change from baseline to after therapy (up to 18 months)
Population: Data was not collected for one participant in the SLIT/OIT A group.
Measure: Median (Full Range); unit: kUa/L
Groups:
- SLIT: These subjects will have a dose escalation of the milk protein extract given sublingually. After dose escalation, they will continue on the sublingual daily maintenance dose for approximately one year.
  Milk Protein Extract Immunotherapy : Sublingual extract daily in escalating doses to goal of 7mg/day for approximately 1 1/2 years.
  Milk Protein Extract Immunotherapy goal of 4mg/day: Sublingual extract given daily in escalating doses with goal of 4 mg/day for approximately 20 weeks.
  Milk Protein Extract Immunotherapy goal of 7mg/day: Sublingual extract daily in escalating doses to goal of 7mg/day for approximately 1 1/2 years.
- SLIT/OIT B: These subjects will start with a dose escalation of the milk protein extract given sublingually, and then will switch to milk powder given orally and will undergo a dose escalation for a goal of 1000 mg. After dose escalation, they will continue on the oral daily maintenance dose for approximately one year.
  Milk Powder Immunotherapy : Milk powder given orally in escalating doses with a goal of 1000mg/day for approximately 1 1/2 years.
  Milk Protein Extract Immunotherapy goal of 4mg/day: Sublingual extract given daily in escalating doses with goal of 4 mg/day for approximately 20 weeks.
  Milk Powder Immunotherapy goal dose 1000mg/day: Milk powder given orally in escalating doses with a goal of 1000mg/day for approximately 1 1/2 years.
- SLIT/ OIT A: These subjects will start with a dose escalation of the milk protein extract given sublingually, and then will switch to milk powder given orally and will undergo a dose escalation for a goal of 2000 mg. After dose escalation, they will continue on the oral daily maintenance dose for approximately one year.
  Milk Powder Immunotherapy : Milk powder given orally in escalating doses with a goal dose of 2000mg/day given for approximately 1 1/2 years.
  Milk Protein Extract Immunotherapy : Sublingual extract given daily in escalating doses with goal of 4 mg/day for approximately 20 weeks.
  Milk Protein Extract Immunotherapy goal of 4mg/day: Sublingual extract given daily in escalating doses with goal of 4 mg/day for approximately 20 weeks.
  Milk Powder Immunotherapy goal dose 2000 mg/day: Milk powder given orally in escalating doses with a goal dose of 2000mg/day given for approximately 1 1/2 years.
Arm/Group | SLIT | SLIT/OIT B | SLIT/ OIT A
Number analyzed (Participants) | 10 | 9 | 9
kUa/L | 0.8 [-390.0 to 10.0] | -13.5 [-170.8 to 471.7] | -9.4 [-49.1 to 42.1]

2. Primary Outcome: Change in CM-specific Immunoglobulin G4 (IgG4)
Description: Cow's milk specific IgG4 was measured at baseline and after therapy (kUa/L)
Time Frame: Change from baseline to after therapy (up to 18 months)
Measure: Median (Full Range); unit: kUa/L
Arm/Group | SLIT | SLIT/OIT B | SLIT/ OIT A
Number analyzed (Participants) | 10 | 10 | 10
kUa/L | 9.9 [0.4 to 705.7] | 157.2 [12.6 to 2415.7] | 31.8 [-16.9 to 798.5]

3. Primary Outcome: Change in End Point Skin Test
Description: Allergen provoked skin test (mm)
Time Frame: Change from baseline to after therapy (up to 18 months)
Measure: Median (Full Range); unit: mm
Arm/Group | SLIT | SLIT/OIT B | SLIT/ OIT A
Number analyzed (Participants) | 10 | 10 | 10
mm | -3.1 [-6.1 to 2] | -3 [-10.9 to 2.3] | -2.5 [-5.1 to 0.9]

4. Primary Outcome: Oral Food Challenge Threshold (OFC) Threshold
Description: mg CM protein
Time Frame: Change from baseline to after therapy (up to 18 months)
Measure: Median (Full Range); unit: mg
Arm/Group | SLIT | SLIT/OIT B | SLIT/ OIT A
Number analyzed (Participants) | 10 | 10 | 10
mg | 2458 [388.9 to 8139] | 8089 [6138.9 to 8130] | 7989 [4289 to 8129]

ADVERSE EVENTS:
Arm/Group | OITA Group | OITB Group | SLIT Group
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OITA Group (N=10) | OITB Group (N=10) | SLIT Group (N=10)
Oropharyngeal inflammation (Gastrointestinal disorders) | 10 (305) | 10 (840) | 10 (1164)

LIMITATIONS AND CAVEATS:
Please refer to the links section, it contains a link to the publication of this research study in the Journal of Allergy and Clinical Immunology

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No